CLINICAL TRIAL: NCT02805738
Title: A Multicenter, Randomized, Double-blind, Parallel Design, Phase III Clinical Trial to Evaluate the Efficacy and Safety of CKD-390 Tablet and Viread® Tablet in Chronic Hepatitis B Patients
Brief Title: Clinical Trial to Evaluate the Efficacy and Safety of CKD-390 Tablet
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 163HBV15036
Record Dates: First submitted 2016-06-16; First posted 2016-06-20 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-04

CONDITIONS: Chronic Hepatitis B
Keywords: Chronic Hepatitis B; tenofovir; CKD-390
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Tenofovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental Group (Experimental): once a time per a day, CKD-390 1 Tablet for each other, PO, During 24 weeks, once a time per a day, 1 tab(CKD-390 1 Tablet) for each other, PO, From 24 weeks to 48 weeks
  Interventions: Drug: CKD-390
- Active comparator Group (Active Comparator): once a time per a day, Viread 1 Tablet for each other, PO, During 24 weeks, once a time per a day, 1 tab(CKD-390 1 Tablet) for each other, PO, From 24 weeks to 48 weeks
  Interventions: Drug: viread

INTERVENTIONS:
Drug: CKD-390 — CKD-390 1 Tablet (48 weeks)
  Other Names: Tenofovir disoproxil aspartate 308.04mg
  Arms: Experimental Group
Drug: viread — viread1 Tablet (24 weeks), CKD-390 1 Tablet (from 24 weeks to 48 weeks)
  Other Names: Tenofovir disoproxil fumarate 300mg
  Arms: Active comparator Group

SUMMARY:
A Multicenter, Randomized, Double-blind, Parallel Design, Phase III Clinical Trial to Evaluate the Efficacy and Safety of CKD-390 tablet

DETAILED DESCRIPTION:
A Multicenter, Randomized, Double-blind, Parallel Design, Phase III Clinical Trial to Evaluate the Efficacy and Safety of CKD-390 tablet and Viread® tablet in Chronic hepatitis B Patients Subjects will receive either a single oral dose of the test formulation(CKD-390) or a oral dose of the reference formulation(viread).

ELIGIBILITY:
Inclusion Criteria:

1. male or female older than 19 years at the time of screening
2. Patients who have chronic hepatitis B disease are taken Viried for 6 months
3. Patients who show HBV DNA undetected(less than 20 IU/mL)
4. Patients who show positive HBsAg
5. Patients who show positive HBeAg or negative HBeAg
6. Patients who fully understand the clinical trials after in-depth explanation, decided to join the clinical trials by their will and signed inform consent

Exclusion Criteria:

1. Patients who are not taken any anti-viral agents except Viread Tab
2. Patients who have hepatitis C (HCV), hepatitis D (HDV), or human immunodeficiency virus (HIV)
3. Patients who have seroperitoneum, icterus, hepatic encephalopathy, variceal hemorrhage or Patients with following value at screening

   * total bilirubin > Upper normal limit x 1.5
   * prothrombin time(INR) > Upper normal limit x 1.5
   * platelets < 75,000/ul
   * serum albumin < 3.0g/dl
4. Patients who are estimated to have hepatocellular carcinoma (HCC) through imaging examination or showed alpha-fetoprotein(AFP) more than 50ng/mL
5. Patients who show Creatinine Clearance < 50 mL/min by calculating Cockcroft-Gault equation
6. Patients with disease like heart failure, renal failure, pancreatitis that investigators consider ineligible for this study
7. Patients who have other hepatic diseases like hematochromatosis, Wilson's disease, alcoholic cirrhosis, autoimmune hepatic diseases, α-1 antitrypsin deficit syndrome
8. Patients with genetic disease like Galactose intolerance, lapplactase deficiency, Glucose-galactose malabsorption
9. History of malignant tumor within 5 years
10. Patients who take any other investigational product within 30 days
11. Patients who have to administer immunosuppressants or Nephrotoxic drugs, Hepatotoxic drugs for period of Clinical Trial
12. Pregnant, breast-feeding and childbearing age who don't use adequate contraception
13. Patients who receive an organ transplant or bone marrow transplant or are going to received surgury
14. History of allergic reaction to the investigational product
15. Patients that investigators consider ineligible for this study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-11 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
The rate of subjects who showed HBV DNA undetected (less than 20IU/mL) | 24weeks after drug administration

SECONDARY OUTCOMES:
The rate of subjects who showed HBV DNA undetected (less than 20IU/mL) | 12, 36, 48 weeks after drug administration
The Difference between the baseline and at the 12, 24, 36, 48 week of HBV DNA level | 12, 24, 36, 48 weeks after drug administration
The rate of subjects who had normal ALT result | 12, 24, 36, 48weeks after drug administration
The rate of subjects who showed HBeAg loss | 24, 48 weeks after drug administration
The rate of subjects who showed HBeAg seroconversion | 24, 48 weeks after drug administration
The rate of subjects who showed HBsAg loss | 24, 48 weeks after drug administration
The rate of subjects who showed HBsAg seroconversion | 24, 48 weeks after drug administration
The rate of subjects who showed Virologic breakthrough | 12, 24, 36, 48 weeks after drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Kwan Sik lee, MD, Principal Investigator — Kangnam severance hospital
Locations (20):
- South Korea (20):
  - Korea University Ansan Hospital, Ansan, Gyeonggi-do
  - Bundang Cha Medical Center, Bundang, Gyeonggi-do
  - Hanyang University Guri Hospital, Guri-si, Gyeonggi-do
  - Inje University Ilsan Paik Hospital, Ilsan, Gyeonggi-do
  - Gachon University of Medicine and Science Gil Medical Center, Incheon, Gyeonggi-do
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Busan National University Hospital, Busan
  - Keimyung University Dongsan Medical Center, Daegu
  - Yeungnam University Medical Center, Daegu
  - Chungnam National University Hospital, Daejeon
  - Jeju National University Hospital, Jeju City
  - Chungang University Hospital, Seoul
  - Hanyang University Hospital, Seoul
  - Kangnam Severance Hospital, Seoul
  - Korea University Guro Hosptial, Seoul
  - Samsung Medical Center, Seoul
  - Seoul Asan Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Seoul Saint Mary's Hospital, Seoul
  - Severance Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No